CLINICAL TRIAL: NCT04383002
Title: Use of High Dose Inhaled Nitric Oxide in Intubated Patients Admitted With COVID-19
Brief Title: High Dose Inhaled Nitric Oxide for COVID-19 (ICU Patients)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-5449
Record Dates: First submitted 2020-05-01; First posted 2020-05-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (control) (No Intervention): Patients will receive standard of care therapy
- Inhaled Nitric Oxide (Experimental)
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — iNO will be given at 160ppm for 6 hours, once a day, for 2 days
  Arms: Inhaled Nitric Oxide

SUMMARY:
Novel therapies are desperately needed for treatment of COVID-19 patients. At present, there are no proven interventions to prevent progression of the disease or to rapidly treat patients with COVID-19 related respiratory failure. Data on the original coronavirus -SARS pneumonia suggested that high dose (>160ppm) inhaled Nitric Oxide could have beneficial effects also on COVID-19, due to the genomic similarities between these two coronaviruses (1-3). This study will test whether high dose inhaled nitric oxide is safe and can reverse virus burden and respiratory failure in patients on mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed infection with COVID-19 positive RT-PCR tracheal aspirate prior to treatment
2. Use of mechanical ventilation with or without ECMO
3. Male or female ages > 18 years
4. < 14 days from symptom initiation to study enrolment and < 7 days from intubation to study enrolment

Exclusion Criteria:

1. Patients on other interventional clinical trials
2. Subjects diagnosed with congestive or unstable heart disease including heart failure, left ventricular dysfunction (LVEF < 40 %) or myocardial damage, severe pulmonary hypertension and/or unstable hypertension
3. Subjects diagnosed with immunodeficiency
4. Hematology: patients with clinically significant anemia e.g. Hemoglobin < 100 and thrombocytopenia e.g. Platelets < 75
5. Subjects with clinically significant history of, or active bleeding including active pulmonary or gastrointestinal bleeding
6. Hepatic Function: Patients with abnormal liver function defined as any two of the following ALT >3x ULN, AST >3x ULN, Total bilirubin < 1.5 X ULN
7. Patient receiving drugs that have a contraindication with NO e.g. use of a nitric oxide donor agent such as nitroglycerin or drugs known to increase methemoglobin such as lidocaine, prilocaine, benzocaine or dapsone at screening as relevant to the proposed study population
8. Pregnancy
9. Subjects with a known hypersensitivity to methylene blue, subjects with glucose-6-phosphate dehydrogenase (G6PD) deficiency
10. Known or suspected thalassemia, sickle cell disease, or other conditions associated with poor oxygen carrying capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
COVID-19 PCR status at completion of treatment (day 7) from tracheal aspirate | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Cypel, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada